CLINICAL TRIAL: NCT00978146
Title: Effect of Hydroxyurea as Treatment for Primary Desmoid Tumors in Adults and Children (CHP-914)
Brief Title: Effect of Hydroxyurea as Treatment for Primary Desmoid Tumors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was administratively withdrawn by the IRB; no subjects were enrolled
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-007317
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Desmoid Tumors; Fibromatosis
MeSH Terms: conditions — Desmoid Tumors; Fibroma | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Desmoid tumor (Experimental): Patients with desmoid tumors
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea — Patients will take oral hydroxyurea with a starting dose of 20 mg/kg daily. Patients will remain on hydroxyurea as long as there is a response or stability in tumor size and associated toxicities are manageable. Maximum treatment duration will be one year.

SUMMARY:
The purpose of this study is to examine the response rate of desmoid tumors to hydroxyurea. The investigators hypothesize that hydroxyurea will be a safe, non-toxic alternative to aggressive surgery or chemotherapy for this difficult to treat tumor.

DETAILED DESCRIPTION:
The treatment of desmoid tumors is complicated by benign histology and potentially aggressive and recurrent behavior. Invasive or intensive treatments with surgery or radiation therapy can lead to good tumor control, but at the expense of significant side effects along with a high risk of local recurrence after surgical excision. Low dose regimens of standard chemotherapy drugs have been favored as a conservative first-line treatment; however, refractory and recurrent tumors are not uncommon. The purpose of this study is to investigate the efficacy and safety of using hydroxyurea, an anti-neoplastic agent with relatively few side-effects, as a novel treatment for primary, unresectable desmoid tumors, desmoid tumors that have had an incomplete primary resection, or desmoid tumors that have recurred after other therapy.

Patients presenting to our oncology center with a new diagnosis of desmoid tumor, or a recurrent desmoid tumor, will be eligible for this study. After informed consent, physical examination, and baseline imaging studies (CT/MRI), patients will receive oral hydroxyurea at a starting dose of 20 mg/kg daily. Laboratory tests will be performed at set intervals to maintain the appropriate dose and monitor for cytopenias. Clinical evaluations, physical examinations, and/or imaging studies will be conducted every three months to assess for changes in tumor size. Patients will remain on hydroxyurea as long as there is a response or stability in tumor size and associated toxicities are manageable. Data will be collected regarding the response to the drug, the duration of the response, and the occurrence of adverse events. The goal of the analysis will be to determine the efficacy of hydroxyurea as a treatment modality for desmoid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients </= 21 years of age will be eligible
* Histologically-confirmed diagnosis of desmoid tumor
* Measurable disease
* Stable hematologic, renal and hepatic parameters
* Negative pregnancy test for women of childbearing potential

Exclusion Criteria:

* Presence of a second neoplastic process
* Pregnant or breastfeeding women, fetuses, and prisoners will not be included in this study
* Patients receiving additional treatment for tumor other than pain control
* Patients having taken an investigational drug within the past 30 days

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of this study is change in tumor size. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Womer, M.D., Study Chair — Children's Hospital of Philadelphia